CLINICAL TRIAL: NCT04640493
Title: The Effect of Sodium Glucose Co-transporter 2 (SGLT2)-Inhibitors on Sleep Disordered Breathing in Heart Failure Patients
Brief Title: SGLT2-Inhibitors for Sleep Apnea in Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAT2147
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Sleep Disordered Breathing
Keywords: heart failure; sleep disordered breathing; sglt2-inhibitor; sglt2; dapagliflozin; watchpat
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Study design is prospective, non-randomized, interventional (non-experimental) pre-post study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SGLT2-SDB (Experimental): Patients with newly diagnosed SDB will be given dapagliflozin (standard dosage, 10mg)
  Interventions: Drug: Dapagliflozin; Device: WatchPat

INTERVENTIONS:
Drug: Dapagliflozin — If patients have been diagnosed with SDB using the WatchPat device, they will start dapagliflozin. Repeat WatchPat SDB assessment will be performed after 3 and 6 months of continuous dapagliflozin therapy.
  Other Names: FARXIGA
Device: WatchPat — HF patients undergo SDB testing with the WatchPat device. (non-experimental)

SUMMARY:
Heart Failure is a disease involving many different aspects of the human body, including changes in metabolism, the way the body produces and uses energy. Research shows that patients with heart failure often have a sleep disorder called sleep disordered breathing (SDB). It has been shown that SDB is associated with poor outcomes in heart failure patients, but the exact reason is unknown. It is likely that SDB leads to changes in metabolism and hormone status in the body, which is especially dangerous for heart failure patients. There is currently no treatment for SDB in heart failure patients. Recently, with Sodium glucose co-transporter 2 (SGLT2)-Inhibitors a new drug class has been approved for the treatment of advanced heart failure. This drug has effects on the metabolism in heart failure patients, among several other effects. This research project has the aim to investigate if SGLT2 inhibitors can help in the treatment of SDB, as many mechanisms of the drug overlap with the mechanisms how SDB develops. The drug has been approved by the FDA for the treatment of heart failure. The investigators want to study the effect of the drug on SDB by using a home sleep test called Watchpat, which has been approved to diagnose SDB.

DETAILED DESCRIPTION:
To explore whether SGLT2-Inhibition has a beneficial effect on Sleep Disordered Breathing (SDB) in advanced heart failure patients. This project proposes to carry out research that addresses the established, but in clinical practice under-recognized association between Sleep Disordered Breathing (SDB) and a worse prognosis in patients with heart failure (HF). SDB is highly prevalent in the HF population. Multiple studies have shown that HF accompanied by SDB is associated with an increased mortality compared to the absence of SDB. Two major types of SDB are prevalent in HF: Obstructive Sleep Apnea (OSA) and Central Sleep Apnea (CSA). Mechanistically, it has been proposed that SDB impacts the neurohumoral axis and systemic metabolism and therefore has particularly detrimental effects on the HF patient population. Therapeutic options for the treatment of SDB are limited. Heart Failure is a multisystemic disease leading to maladaptive cardiac and systemic metabolic changes. Recently, with SGLT2-Inhibitors a new drug class has been approved for the treatment of advanced heart failure. This is the first drug class in the HF drug armamentarium targeting cardiometabolic mechanisms. This study seeks to improve the health of individuals with heart failure by exploring whether SGLT2-Inhibition has a beneficial effect on SDB (OSA and CSA) in advanced heart failure patients and therefore may be a novel therapeutic option for the treatment of SDB in advanced HF. The specific aim of this project is to assess the effect of therapy with a SGLT2-I on SDB in ambulatory advanced HF patients by using the WatchPAT-derived apnea-hypopnea index as well as subjective measures of sleep quality using the Berlin Questionnaire and Epworth Sleepiness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Consent-able adults
* Diagnosis of heart failure
* Diagnosis of SDB
* No contraindication for taking dapagliflozin

Exclusion Criteria:

* Patients without heart failure
* Patients without SDB
* Contraindication for taking dapagliflozin (severe renal impairment, hemodialysis, or history of severe hypoglycemic episodes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea Index | 6 months
  Change in the apnea-hypopnea index as measured by the WatchPAT device.
Change Berlin Questionnaire Categorization | 6 months
  The Berlin Questionnaire for sleep apnea consists of 3 categories related to the risk of having sleep apnea. Participants are classified as "High Risk" or "Low Risk" for sleep apnea. High risk categorization is assigned when there are 2 or more categories where the score is positive ("positive" defined as a score of 2 or more points). Low risk categorization is assigned when there is 1 or no categories where the score is positive.
Change in Epworth Sleepiness Scale | 6 months
  The Epworth Sleepiness Scale is an 8-item scale measuring sleepiness in various situations. Each situation is scored as 0=no chance of dozing to 3= high chance of dosing. Scores range from 0-24, with a higher score indicating a higher level of sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Uriel, MD, Principal Investigator — Columbia University
Locations (1):
- Vivian and Seymour Milstein Family Heart Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No